CLINICAL TRIAL: NCT06804668
Title: Safety and Feasibility of Tele-supervised Home-based Transcranial Direct Current Stimulation in Parkinson's Disease
Acronym: Home-PD-tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Michael D. Fox, M.D.,Ph.D., Director, Center for Brain Circuit Therapeutics, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2024P001978
Record Dates: First submitted 2025-01-22; First posted 2025-02-03 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Brain stimulation; Parkinson; Movement disorder; Non-invasive brain stimulation
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Masking Description: Scores will be recorded on video to ensure blinding to the timepoint of clinical scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Active tDCS (Experimental): Subjects receiving active tDCS
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — The intervention involves a home-based, self-administered application of network-targeted, multifocal transcranial direct current stimulation (tDCS) using the Neuroelectrics® StarStim Home-tES device. Participants will apply the tDCS for 20 minutes each day over seven consecutive days. The device is specifically programmed to target a brain network associated with motor symptom improvement in Parkinson's Disease, based on recent research identifying this network through deep brain stimulation studies.

SUMMARY:
The goal of this clinical trial is to learn whether home-based transcranial direct current stimulation (tDCS) is safe and practical for people aged 40 to 70 years with Parkinson's Disease. The study aims to find out if participants can use the tDCS device at home without serious side effects and whether it is easy for them to use on their own.

Participants will first attend an in-person visit to learn how to use the tDCS device. They will then use the device at home once a day for 20 minutes over seven consecutive days. Video calls on days 2 and 3 will provide support and supervision. After each session, participants will complete brief online questionnaires about any side effects and how easy the device was to use. The study will also check if using tDCS at home improves motor symptoms in Parkinson's Disease by using a standard movement assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of Parkinson's disease, aged between 40 and 70, who provide verbal and written informed consent will be included. Patients should have access to a computer system for video calls and completing the questionnaires, and they must be able to use it.

Exclusion Criteria:

* Psychiatric symptoms such as moderate or severe depression
* Cranial metal implants
* Cardiac pacemaker
* Epilepsy, stroke
* Substance abuse
* Inability to adjust the neoprene cap with the electrodes independently due to movement disturbances

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of repeated network-targeted multifocal tDCS at home | 8 days.
  Measures the total number of days each participant successfully completes tDCS sessions at home, aiming for seven consecutive days.
  Method:
  Daily online logs.

SECONDARY OUTCOMES:
Safety of repeated network-targeted multifocal tDCS at home | 8 days.
  Counts adverse events related to tDCS or technical difficulties over the 8-day period.
Questionnaires for difficulty in usability, subjective effect on motor symptoms, severity of side effects | 8 days.
  Visual analogue scales (VAS, 0-10) will be performed daily. 0 is the minimum and 10 the maximum score.
Motor outcome | 8 days.
  Outcome in MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS). This score is specifically designed to assess the motor symptoms of Parkinson's disease.
  Scoring Range:
  * Minimum Score: 0 (No motor impairment)
  * Maximum Score: 132 (Severe motor impairment)

OTHER OUTCOMES:
Support | 8 days.
  Open point: level and amount of support needed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Fox, MD, PhD, Principal Investigator — Center for Brain Circuit Therapeutics, Department of Neurology, Brigham & Women's Hospital, Boston, MA
Locations (1):
- Center for Brain Circuit Therapeutics, Department of Neurology, Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data collected during the study after de-identification (removal of personal identifiers).
  Data to be Shared:
  * De-identified individual participant data, including:
  * Demographic information (age range, gender)
  * Clinical assessments such as MDS-UPDRS-III scores
  * Responses to usability and side effect questionnaires
  * Information on any reported adverse events
Supporting Information: Study Protocol